CLINICAL TRIAL: NCT03280329
Title: Music Therapy in the ICU as a Tool to Reduce Neuroactive Drugs: Generalized Versus Personalized Intervention
Brief Title: Generalized Versus Personalized Music Therapy in the ICU to Reduce Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giovanni Mistraletti, University researcher, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Musicoterapia
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Critical Illness; Hypnotics and Sedatives; Music Therapy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): the patients who belong to this group will not be assigned to a regulated music therapy treatment, thus they will listen to the background sounds (alerts, voices) right in the Intensive Care environment; radio use will be allowed according to medical/ nursing judgements
- Personalised treatment (Active Comparator): A music therapy advice will be performed with each patient (if possible from the neurological point of view) or their caregivers to assess their musical preferences and a list of songs will be generated which will be reproduced for 2 hours per day from admission to discharge with the use of earphones.
  Interventions: Other: Personalized Music therapy
- Generalized treatment (Active Comparator): Music will be broadcasted in each patient room after the creation of a 'weekly playlist' with the following considerations:
  1. Daily sound reproduction from 7 am to 11 pm, with 10 minutes break about every 50 minutes of music;
  2. Spread through the environment with specifically designated speakers, at a controlled volume (30-50 dB);
  3. Choice of playlist of music both classic and modern, with very easy listening, selected according to the daily hours to restore circadian rhythm and following predictable activities of care provided to patients (hygienic care, retail food, administration other therapies, physiotherapy, visit by relatives, …);
  4. Mixing tracks so that there is continuity and fluidity of listening
  Interventions: Other: Generalized Music therapy

INTERVENTIONS:
Other: Generalized Music therapy — Patients will receive broadcasted music via speakers in their room from 7am to 11pm, from admission to discharge
  Arms: Generalized treatment
Other: Personalized Music therapy — Patients will receive music via earphones after specific music therapist advice, for 2 hours per day, from admission to discharge
  Arms: Personalised treatment

SUMMARY:
Admission to an Intensive Care Unit (ICU) is one of the major causes of stress and both physical and emotional difficulties for critically ill patients, both because of the illness that caused the admission and of the ICU nevironment itself. Despite the use of protocols and tools to evaluate sedation, many patients continue to have high levels of anxiety. An inadequate treatment of this condition is associated with increased sympathetic activity which causes dyspnea and an increase in myocardial oxygen consumption. Sedative drugs, on the other side, may have significant side effects.

In view of this, there is clear need to find new strategies and instruments allowing for the maximization of critical patients' comfort, by promoting pain, anxiety, stress and agitation relief and minimising the need of sedative therapy.

The main hypothesis of this study is that the use of music therapy for critically ill patients can lead to a significant increase of the days free from neuroactive therapy (analgesics, sedatives, antianxiety meds, antipsychotics) in the first 28 days following Intensive Care Unit admission. To this purpose, data obtained from 3 groups of patients will be compared - a group with individual treatment administered by a music therapist and delivered by headphones, a group with a generalised treatment, through the creation of a weekly musical program continuously broadcasted in the hospital room, and a control group.

DETAILED DESCRIPTION:
Introduction The Intensive Care Unit (ICU) is one of the major causes of stress and both physical and emotional difficulties for patients and their families.

Studies have been conducted in the investigators' and other Intensive Care Units and they set out to investigate main causes of stress in critical patients; among the most significant factors were shown to be life saving treatment such as mechanical ventilation, invasive procedures, restriction of movement, pain and inability to verbally express it, environment characterized by constant light and sound stimulation, loss of interaction with loved ones and the staff, and sleep deprivation.

Despite the use of protocols and tools to evaluate sedation, many patients continue to have high levels of anxiety. An inadequate treatment of this condition is associated with increased sympathetic activity which causes dyspnea and an increase in myocardial oxygen consumption.

In view of it, there is clear need to find new strategies and instruments allowing for the maximization of critical patients' comfort, by promoting pain, anxiety, stress and agitation relief and minimising the need of sedative therapy.

Among non pharmacological treatment, hypnosis and relaxation techniques, implementation of communication with patient, music therapy and physical support are shown to be effective (7).

The use of music as a therapeutic complement has been described in literature for a long time, using a rational selection in musical composition. Music application to obtain health benefit is defined music therapy.

The main research question which this study aims to answers is music therapy's effectiveness in reducing analgesics and sedatives need, as well as reducing anxiety and loneliness, and in re- establishing normal sleep patterns. It should be noted that music brings significant benefits as there is absence of contraindications and it is immediately usable by everybody. Italian experiences in the music therapy field in the Intensive Care Unit are low.

With this music therapy project, the investigators intend to build a multifactorial intervention to reduce stress risk factors of patients and their families, still not applied in our country.

Rationale

Many factors influence the effectiveness by music therapy: age, gender, cognitive abilities, stress levels, anxiety, pain, music education, familiarity with a determinate type of music, individual preferences, and culture are all elements which can modify the effect of certain music selection on the subject (19, 20). From this, there is the need of individual choice and careful monitoring of effects that music has on each individual.

Music therapy in the treatment of stress in the Intensive Care Unit

A recent meta analysis (21) reveals that listening to music can cause a reduction of anxiety levels in mechanically ventilated patients; some studies show, moreover, a reduction of analgesic and sedative need in response to the application of a music therapy treatment.

Mechanisms underlying music therapy effectiveness A shared theory about the reduction of anxiety induced by music is that it helps patients to distance their minds from environmental stress factors to focus on pleasant sounds and calming incentives (8, 22).

The effect of music is extensive, moreover giving patients an aesthetic experience which offers comfort and peace in a stressful situation. Guided interventions by music therapists are more effective because music used is adapted to the needs of that determinate moment, thanks to professional abilities. If music is selected personally by patient, this provides a major sense of control in the environment, like that of Intensive Unit, where the patient is almost totally dependent from health workers (23).

From the neuropsychological point of view, it was assumed that music has a relaxing effect through its impact on central and autonomic nervous system (24- 26); more specifically, its application determines a deleting effect on the sympathetic system, leading to a reduction of circulating catecholamines and to lower nervous and muscle stimulation (25,27). Potential benefits which result are reduction of pain, reduction of blood pressure, heart rate, oxygen consumption and muscle tension (2).

Hypothesis of the study The hypothesis of this study is that the use of music therapy for critically ill patients can lead to a significant increase of the days free from neuroactive therapy (analgesics, sedatives, antianxiety meds, antipsychotics) in the first 28 days following Intensive Care Unit admission, in absence of statistically significant reduction of the welfare index of health workers.

All these data are not available in the literature and would represent an undiscussed advantage in the promotion of welfare in critical patients during recovery in Intensive Care and at distance from itself; this can also lead to possible significant implications in terms of a more effective assistance and lower duration of the stay.

Purpose of the study

The present study study has the main purpose of verifying if using music therapy as an individualised or generalized intervention in hospitalised patients in Intensive Care, in different cure settings, allows for a reduction of total dose of analgesics/sedatives/antipsychotics administered. The investigators will analyse if the proposed intervention of music therapy can have a role in giving the following advantages:

* increased hours of sleep of patients,
* reduction of anxiety and psychomotor agitation manifestations,
* improvement of work welfare,
* lower grade of anxiety, stress, and post traumatic symptoms of the family,
* reduction of frequency and duration of physical restraint,
* practicability of the proposal of generalized music therapy, through the understanding the frequency in which music is interrupted for reasons of clinical contingency.

To this purpose, data obtained from 3 groups of patients will be compared - a group with individual treatment, a group with generalised treatment, through the creation of a weekly musical program, and a control group.

The population in study will be that of patients hospitalised in Intensive Care for variable aetiologies, which recovery is longer than 3 days.

All without undermine (or even improve) worker welfare, in order to improve physical and psychological outcome of patients.

Protocol

Randomization and study groups

The 3 groups are:

1. Control: the patients who belong to this group will not be assigned to a regulated music therapy treatment, thus they will listen to the background sounds (alerts, voices) right in the Intensive Care environment; radio use will be allowed according to medical/ nursing judgements;
2. Personalised treatment: during a music therapy consultancy, each patient will be investigated (if possible from the neurological point of view) on musical preferences and list of possible music will be proposed which will be reproduced for 2 hours at day. It is specified that this genre of intervention, as far as well described and studied in literature, does not belong in clinical practice, and therefore earphones for listening to music are not yet used in our task force.
3. Generalised treatment: it will be carried out through the creation of a 'weekly playlist' with the following considerations:

   1. Daily sound reproduction from 7 am to 11 pm, with 10 minutes break about every 50 minutes of music;
   2. Spread through the environment with specifically designated speakers, at a controlled volume (30-50 dB);
   3. Choice of playlist of music both classic and modern, with very easy listening, selected according to the daily hours to restore circadian rhythm and following predictable activities of care provided to patients (hygienic care, retail food, administration other therapies, physiotherapy, visit by relatives, …);
   4. Mixing tracks so that there is continuity and fluidity of listening.

Patients will be randomly assigned to the study groups. On the basis that proposed intervention has environmental nature (in control and music therapy group), patients respecting inclusion and exclusion criteria to the protocol will be divided according to the room occupied. The study is configured like a randomized study, not a blind one.

The environment where the study will take place, the departement of Anestesia e Rianimazione of San Paolo Hospital - University, does not have single box but 3 open rooms, each one with 2 beds, in which single beds are separated by about 5 meters. This logistic issue will not hinder the study execution since nothing changes with control group patients about sound environmental management; for personalized music therapy group the use of earphones avoid the music overlap coming from the other patients; equally for the generalized music therapy, in view of intervention nature which provides passive exposure of patients to the music reproduced in the whole environment of the room, the results will not be relatively impacted by the ward. The 3 rooms are instead well disjoint among themselves, so that music coming from one hardly can reach the others.

Collected data It will be measured for each patient's' free days from neuroactive drugs and neuroactive drug total dosage administered. Moreover, the eventual need of use of restraints for patient safety and duration will be registered.

Once per nursing shift, anxiety levels will be detected, measured with verbal scale number (VNR), agitation, measured with RASS scale (Richmond Agitation- Sedation Scale), and pain will be detected with VNR scale or behavioural measures (Behavioral Pain Scale, BPS).

Moreover the hours of sleep declared in medical record will be registered on the basis of nurse evaluations.

Through semi structured interviews, welfare of the health care workers and relatives will be investigated as well as the perceived interference of the intervention based on music therapy; the impact of experience in Intensive Care on the lives of relatives will be evaluated through a validated questionnaire (SSS- Short Scale for PTSS).

In order to verify the feasibility of the proposal of generalised music therapy, the number of interruptions of music reproduction will be registered for contingent clinical reasons.

Analysis of data From the data collected, organised in a database in compliance with the applicable privacy policy (law 196/2003), it will be possible to verify if the use of personalised and generalised music therapy in patients hospitalized in Intensive Care, in different care settings, allows for a reduction of total dosage of analgesic/ sedative/ antipsychotic drugs administered.

All the analysis will be centralised at the investigators' institution.

Sample size Assuming the possibility to transform data with Blom method, in order to obtain a normal distribution and so higher power in equal amplitude sample, and assuming a effect size of 0.30 and a doubling of the parameter of main outcome (days free from neuroactive drugs administration) in the 2 groups of intervention compared to the control group, the sample size required or an effective power of 80% is 53 subjects per group. This sample size is also sufficient to cover the analysis conducted comparing measurements repeated on the same patient. To this purpose, a linear model will be used which requires 51 subjects per groups, assuming a correlation coefficient of 0.5 between measures and a size effect of 0.25. Sizing was conducted with SAS software.

Statistical analysis Data will be expressed as median (standard deviation) if normally distributed (Shapiro- Francia test), or like median ( range interquartile) otherwise. Data will be transcribed from clinical records on a sheet of Microsoft Excel 2010 calculations (Microsoft Corporation, Redmond, WA, USA). Statistical analysis will be performed with Stata/SE 12.0 (StataCorp, College Station, TX USA). For each comparison statistical significance will be considered for values of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized in Intensive Care for any medical, surgical traumatic condition, whose stay in the ICU is expected to be longer than 2 days

Exclusion Criteria:

* expected Glascow Goma Scale at ICU discharge lower than 12
* hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Neuroactive drug free days | one year
  the outcome will be calculated giving one point for each day during the measurement period that patients are both alive and free the administration of any neuroactive drug

SECONDARY OUTCOMES:
Sedative exposure | one year
  Sedative exposure will be determined for all patients who will receivd any of 8 commonly administered sedative and analgesic medications in the ICU (midazolam, lorazepam, propofol, dexmedetomidine, morphine, fentanyl, hydromorphone, haloperidol) 24 hours prior to enrollment and each day during the study. Sedative exposure will be operationalized as a daily sedative drug intensity score and sedative dose frequency
reduction of the stress associated to ICU stay | one year
  the stress during the ICU stay will be measured by the validated ICUESS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo - Polo Universitario, Milan, Italy

REFERENCES:
- [Derived] Mistraletti G, Solinas A, Del Negro S, Moreschi C, Terzoni S, Ferrara P, Negri K, Calabretta D, Formenti P, Formenti A, Umbrello M. Generalized music therapy to reduce neuroactive drug needs in critically ill patients. Study protocol for a randomized trial. Trials. 2024 Jun 12;25(1):379. doi: 10.1186/s13063-024-08220-8. PMID 38867317